CLINICAL TRIAL: NCT03005041
Title: A Clinical Study Evaluating the Consumer Perception of an Experimental Mouthwash Formulation After a Single Use
Brief Title: Consumer Perception of an Experimental Mouthwash After a Single Use in Dry Mouth Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 205067
Record Dates: First submitted 2016-08-30; First posted 2016-12-29 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-08

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product 1 (Experimental): Participants will rinse their mouth with 15 mL of the product swishing for 30 seconds.
  Interventions: Other: Biotene mouthwash
- Test Product 2 (Other): Participants will rinse their mouth with 15 mL of the water swishing for 30 seconds. Participants then spit out the water.
  Interventions: Other: Bottled mineral water

INTERVENTIONS:
Other: Biotene mouthwash — Participants will rinse their mouth with 15 mL of Biotene mouthwash swishing for 30 seconds.
  Arms: Test Product 1
Other: Bottled mineral water — Participants will rinse their mouth with 15 mL of the water swishing for 30 seconds.
  Arms: Test Product 2

SUMMARY:
The purpose of this study is to investigate the consumer perception of an experimental mouthwash formulation in population with dry mouth

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Aged 18 - 84 years inclusive
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon oral examination
* Participant reports having a feeling of a dry mouth according to the Dry Mouth Screening Questionnaire (DMSQ) (Subject must answer at least 2 out of the 4 questions with 'agree a little', 'agree' or 'strongly agree' at the Screening Visit (Visit 1). Participants with un-stimulated whole salivary flow rate of ≤0.1 ml/min at the Screening Visit (Visit 1).
* Participants with un-stimulated whole salivary flow rate of ≤0.1 ml/min ATH the Screening Visit (Visit 1).
* Understands and is willing, able and likely to comply with all study procedures and restrictions

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study or have a positive urine pregnancy test at the Screening Visit
* Women who are breast-feeding
* Participant is currently undergoing radiotherapy and/or chemotherapy treatment
* Any condition the investigator identifies that can confound the participant's ability to properly participate in the study e.g. Alzheimer's Disease
* Participant with untreated oral mucosal disease which in the opinion of the investigator could interfere with the study (e.g. current oral ulceration)
* Evidence of gross intra-oral neglect or need for extensive dental therapy
* Denture wearer (complete dentures)
* Participant not on stable doses of prescription systemic parasympathetic medications (e.g. Pilocarpine), for the treatment of the feeling of dry mouth
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 14 days of the screening visit
* Previous participation in this study
* Recent history (within the last 1 year) of alcohol or other substance abuse
* An employee of the sponsor or the clinical study team or members of their immediate family. Students and employees of the Tufts University School of Dental Medicine not associated with the clinical trials team are eligible to participate. Students and employees will not be specifically targeted for enrollment
* Non-English speaking Participants will not be enrolled in the study. Participants must be able to read and write in English

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single center in United states of America (U.S.A)
Pre-assignment Details: A total 58 participants were screened, out of which 56 participants were enrolled in the study. Two participants were not enrolled as they did not meet the study criteria. Of 56 enrolled participants, 55 participants were randomized as one participant withdrew consent.
Groups:
- Experimental Oral Rinse/Mineral Water: Participants were supervised to rinse their mouth with 15 milliliter (mL) of the experimental oral rinse/mouth wash swishing followed by with 15mL of mineral water swishing in period 1 and period 2 respectively. Participants then spat out products after rinsing for 30 seconds. No rinsing with water immediately after experimental oral rinse/mouth wash use was permitted. Each period was separated by a washout period of minimum 24 hours to maximum 7 days.
- Mineral Water/Experimental Oral Rinse: Participants were supervised to rinse their mouth with 15 mL of the mineral water swishing followed by with 15mL of experimental oral rinse/mouth wash swishing in period 1 and period 2 respectively. Participants then spat out products after rinsing for 30 seconds. No rinsing with water immediately after experimental oral rinse/mouth wash use was permitted. Each period was separated by a washout period of minimum 24 hours to maximum 7 days.
Period: Period 1
Arm/Group | Experimental Oral Rinse/Mineral Water | Mineral Water/Experimental Oral Rinse
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0
Period: Washout Period 1
Arm/Group | Experimental Oral Rinse/Mineral Water | Mineral Water/Experimental Oral Rinse
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Experimental Oral Rinse/Mineral Water | Mineral Water/Experimental Oral Rinse
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Participants: All randomized participants who received both the treatments experimental oral rinse/mouthwash and mineral water were included in the baseline assessment.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response to Post-Product Use Questionnaires 1 (PPUQ 1); Question No.1
Description: Participants answered the following question, Q1: how much do you agree or disagree with the following statements about this product, having used it? "This product is gentle": disagree strongly, disagree, neither agree nor disagree, agree, or agree strongly. There was no formal statistical hypothesis to be tested for this outcome..
Time Frame: Within 2 minutes post product use
Population: Analysis for this outcome was performed on intent to treat (ITT) population which included all the participants who were randomized, received at least one dose of treatment during the study and had at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental Oral Rinse: Participants were supervised to rinse their mouth with 15 mL of the experimental oral rinse/mouth wash swishing for 30 seconds. Participants then spat out product. No rinsing with water immediately after experimental oral rinse/mouth wash use was permitted.
- Mineral Water: Participants were supervised to rinse their mouth with 15 mL of the mineral water swishing for 30 seconds. Participants then spat out the water.
Arm/Group | Experimental Oral Rinse | Mineral Water
Number analyzed (Participants) | 55 | 55
Participants
  Disagree Strongly | 1 | 1
  Disagree | 5 | 0
  Neither Agree nor Disagree | 6 | 5
  Agree | 26 | 21
  Agree Strongly | 17 | 28

2. Secondary Outcome: Number of Participants With Response to Post-Product Use Questionnaires 1 (PPUQ 1); Question No. 3-7
Description: Participants answered the following questions, Q3: Which of following statements best describes how much you liked product overall? liked it-extremely, very much, somewhat, slightly, did not like it that much, did not like it at all. Q 4: Which of the following statements best describes how much you liked overall flavor of rinse? liked it-extremely, very much, somewhat, slightly, did not like it that much, did not like it at all. Q 5: How you would rate flavor intensity of oral rinse? strongest flavor imaginable, very strong, strong, moderate, weak, barely detectable, no flavor at all. Q 6: Did you experience any of following sensations in your mouth & how strong was sensation? moisturizing, soothing, refreshing, tingling, numbing, burning, or drying out. Participants who selected "None" for a particular sensation, did not complete Q 7 for that sensation: When did you experience sensations in your mouth? initially, during use, or after use.
Time Frame: Within 2 minutes post product use
Population: ITT population which included all the participants who were randomized, received at least one dose of treatment during the study and had at least one post-baseline assessment. Note: Number of participants who answered question 6 proceeded to answer question 7. Participants also chosen more than one answer for question 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Oral Rinse | Mineral Water
Number analyzed (Participants) | 55 | 55
Participants
  Q3: Liked it extremely | 13 | 7
  Q3: Liked it very much | 27 | 15
  Q3: Liked it somewhat | 4 | 13
  Q3: Liked it slightly | 6 | 9
  Q3: Did not like it that much | 4 | 7
  Q3: Did not Like it at all | 1 | 4
  Q4: Liked it extremely | 16 | 9
  Q4: Liked it very much | 18 | 9
  Q4: Liked it somewhat | 8 | 14
  Q4: Liked it slightly | 8 | 7
  Q4: Did not like it that much | 3 | 11
  Q4: Did not Like it at all | 2 | 5
  Q5: Strongest flavor imaginable | 5 | 0
  Q5: Very strong | 4 | 1
  Q5: Strong | 19 | 0
  Q5: Moderate | 27 | 6
  Q5: Weak | 0 | 4
  Q5: Barely detectable | 0 | 11
  Q5: No flavor at all | 0 | 33
  Q6(Moisturizing): None | 3 | 12
  Q6(Moisturizing): Mild | 12 | 21
  Q6(Moisturizing): Moderate | 30 | 20
  Q6(Moisturizing): Severe | 10 | 2
  Q7(Moisturizing)Initially-first contact with mouth: number analyzed (Participants) | 52 | 43
  Q7(Moisturizing)Initially-first contact with mouth | 30 | 30
  Q7Moisturizing:During use-whilst swishing in mouth: number analyzed (Participants) | 52 | 43
  Q7Moisturizing:During use-whilst swishing in mouth | 30 | 27
  Q7Moisturizing:After use-spitting out product: number analyzed (Participants) | 52 | 43
  Q7Moisturizing:After use-spitting out product | 34 | 17
  Q6(Soothing): None | 3 | 15
  Q6(Soothing): Mild | 11 | 18
  Q6(Soothing): Moderate | 28 | 19
  Q6(Soothing): Severe | 13 | 3
  Q7(Soothing): Initially - first contact with mouth: number analyzed (Participants) | 52 | 40
  Q7(Soothing): Initially - first contact with mouth | 23 | 22
  Q7(Soothing): During use -whilst swishing in mouth: number analyzed (Participants) | 52 | 40
  Q7(Soothing): During use -whilst swishing in mouth | 34 | 30
  Q7(Soothing):After use-after spitting out product: number analyzed (Participants) | 52 | 40
  Q7(Soothing):After use-after spitting out product | 28 | 11
  Q6(Refreshing): None | 3 | 15
  Q6(Refreshing): Mild | 7 | 19
  Q6(Refreshing): Moderate | 27 | 19
  Q6(Refreshing): Severe | 18 | 1
  Q6(Refreshing): Missing | 0 | 1
  Q7(Refreshing): Initially-first contact with mouth: number analyzed (Participants) | 52 | 39
  Q7(Refreshing): Initially-first contact with mouth | 30 | 20
  Q7(Refreshing):During use-whilst swishing in mouth: number analyzed (Participants) | 52 | 39
  Q7(Refreshing):During use-whilst swishing in mouth | 32 | 22
  Q7(Refreshing)After use-after spitting out product: number analyzed (Participants) | 52 | 39
  Q7(Refreshing)After use-after spitting out product | 32 | 13
  Q6(Tingling): None | 24 | 48
  Q6(Tingling): Mild | 13 | 4
  Q6(Tingling): Moderate | 14 | 1
  Q6(Tingling): Severe | 3 | 0
  Q6(Tingling): Missing | 1 | 2
  Q7(Tingling): Initially-first contact with mouth: number analyzed (Participants) | 30 | 5
  Q7(Tingling): Initially-first contact with mouth | 10 | 0
  Q7(Tingling):During use - whilst swishing in mouth: number analyzed (Participants) | 30 | 5
  Q7(Tingling):During use - whilst swishing in mouth | 17 | 4
  Q7(Tingling):After use -after spitting out product: number analyzed (Participants) | 30 | 5
  Q7(Tingling):After use -after spitting out product | 12 | 1
  Q6(Numbing): None | 44 | 52
  Q6(Numbing): Mild | 8 | 0
  Q6(Numbing): Moderate | 2 | 1
  Q6(Numbing): Severe | 0 | 0
  Q6(Numbing): Missing | 1 | 2
  Q7(Numbing): Initially-first contact with mouth: number analyzed (Participants) | 10 | 1
  Q7(Numbing): Initially-first contact with mouth | 3 | 1
  Q7(Numbing):During use - whilst swishing in mouth: number analyzed (Participants) | 10 | 1
  Q7(Numbing):During use - whilst swishing in mouth | 2 | 1
  Q7(Numbing):After use - after spitting out product: number analyzed (Participants) | 10 | 1
  Q7(Numbing):After use - after spitting out product | 4 | 0
  Q6(Burning): None | 45 | 53
  Q6(Burning): Mild | 5 | 0
  Q6(Burning): Moderate | 2 | 0
  Q6(Burning): Severe | 2 | 0
  Q6(Burning): Missing | 1 | 2
  Q7(Burning): Initially-first contact with mouth: number analyzed (Participants) | 9 | 0
  Q7(Burning): Initially-first contact with mouth | 2 | 0
  Q7(Burning):During use - whilst swishing in mouth: number analyzed (Participants) | 9 | 0
  Q7(Burning):During use - whilst swishing in mouth | 4 | 0
  Q7(Burning):After use - after spitting out product: number analyzed (Participants) | 9 | 0
  Q7(Burning):After use - after spitting out product | 3 | 0
  Q6(Drying Out): None | 49 | 47
  Q6(Drying Out): Mild | 4 | 3
  Q6(Drying Out): Moderate | 1 | 1
  Q6(Drying Out): Severe | 0 | 2
  Q6(Drying Out): Missing | 1 | 2
  Q7(Drying Out): Initially-first contact with mouth: number analyzed (Participants) | 5 | 6
  Q7(Drying Out): Initially-first contact with mouth | 1 | 2
  Q7(Drying Out):During use-whilst swishing in mouth: number analyzed (Participants) | 5 | 6
  Q7(Drying Out):During use-whilst swishing in mouth | 1 | 1
  Q7(Drying Out)After use-after spitting out product: number analyzed (Participants) | 5 | 6
  Q7(Drying Out)After use-after spitting out product | 5 | 4

3. Secondary Outcome: Number of Participants With Response to Post-Product Use Questionnaires 2 (PPUQ 2)
Description: Participants answered the following question; Q1: Are you experiencing any of the following sensations in your mouth and how strong is the sensation? moisturizing, soothing, refreshing, tingling, numbing, burning, or drying out. Q2: Would you continue use of the product? (Yes or No)
Time Frame: Within 30 ± 5 minutes post product use
Population: Analysis for this outcome was performed on ITT population which included all the participants who were randomized, received at least one dose of treatment during the study and had at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Oral Rinse | Mineral Water
Number analyzed (Participants) | 55 | 55
Participants
  Q1: Moisturizing: None | 7 | 27
  Q1: Moisturizing: Mild | 20 | 22
  Q1: Moisturizing: Moderate | 23 | 5
  Q1: Moisturizing: Severe | 5 | 1
  Q1: Soothing: None | 9 | 35
  Q1: Soothing: Mild | 20 | 14
  Q1: Soothing: Moderate | 24 | 3
  Q1: Soothing: Severe | 2 | 1
  Q1: Soothing: Missing | 0 | 2
  Q1: Refreshing: None | 10 | 38
  Q1: Refreshing: Mild | 24 | 7
  Q1: Refreshing: Moderate | 17 | 6
  Q1: Refreshing: Severe | 4 | 1
  Q1: Refreshing: Missing | 0 | 3
  Q1: Tingling: None | 46 | 51
  Q1: Tingling: Mild | 7 | 1
  Q1: Tingling: Moderate | 2 | 0
  Q1: Tingling: Severe | 0 | 0
  Q1: Tingling: Missing | 0 | 3
  Q1: Numbing: None | 52 | 50
  Q1: Numbing: Mild | 2 | 2
  Q1: Numbing: Moderate | 1 | 1
  Q1: Numbing: Severe | 0 | 0
  Q1: Numbing: Missing | 0 | 2
  Q1: Burning: None | 53 | 51
  Q1: Burning: Mild | 1 | 0
  Q1: Burning: Moderate | 0 | 1
  Q1: Burning: Severe | 0 | 1
  Q1: Burning: Missing | 1 | 2
  Q1: Drying Out: None | 45 | 36
  Q1: Drying Out: Mild | 6 | 5
  Q1: Drying Out: Moderate | 1 | 5
  Q1: Drying Out: Severe | 2 | 7
  Q1: Drying Out: Missing | 1 | 2
  Q2: Would You Continue Use of The Product? Yes | 43 | 20
  Q2: Would You Continue Use of The Product? No | 12 | 35

4. Secondary Outcome: Number of Participants With Response to Product Performance Attribute Questionnaire (PPAQ)
Description: Participants rated the following criteria on a scale of 1 to 5(1=Poor, 2= Fair, 3= Good, 4= Very good, 5= Excellent) as follows: 1. Having an immediate dry mouth relief, 2. Having an immediate lubricating effect, 3. Having an immediate moisturizing effect.
Time Frame: Within 5 minutes post product use
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Oral Rinse | Mineral Water
Number analyzed (Participants) | 55 | 55
Participants
  Q1: Excellent | 14 | 4
  Q1: Very good | 22 | 9
  Q1: Good | 7 | 19
  Q1: Fair | 9 | 13
  Q1: Poor | 3 | 10
  Q2: Excellent | 13 | 2
  Q2: Very good | 19 | 9
  Q2: Good | 10 | 13
  Q2: Fair | 11 | 16
  Q2: Poor | 2 | 15
  Q3: Excellent | 13 | 3
  Q3: Very good | 21 | 7
  Q3: Good | 9 | 18
  Q3: Fair | 11 | 13
  Q3: Poor | 1 | 14

ADVERSE EVENTS:
Groups:
- Experimental Oral Rinse: Participants were supervised to rinse their mouth with 15 mL of the experimental oral rinse/mouth wash swishing for 30 seconds. Participants then spat out product. No rinsing with water immediately after experimental mouth wash use was permitted.
Arm/Group | Experimental Oral Rinse | Mineral Water
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 1/55 | 0/55
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Oral Rinse (N=55) | Mineral Water (N=55)
Cyst (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.